CLINICAL TRIAL: NCT04095013
Title: Comparative Evaluation of Intrathecal Bupivacaine-fentanyl and Bupivacaine-dexmedetomidine for Elective Low Segment Caesarean Section
Brief Title: Intrathecal Bupivacaine-fentanyl and Bupivacaine-dexmedetomidine for Elective Low Segment Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sana Urooj, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: dr.sanaurooj@yahoo.com
Record Dates: First submitted 2019-09-14; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Cesarean Section Complications
Keywords: Elective low segment caesarean section; Intrathecal; bupivacaine-fentanyl; bupivacaine-dexmedetomidine; sensory block; complications; hemodynamics
MeSH Terms: interventions — Bupivacaine; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomize controlled trial (RCT)
Who Masked: Participant, Care Provider
Masking Description: Patients were randomly allocated into two groups and will be blinded to the study drugs. The drugs will be chosen by seal envelope method by principal investigator and co-investigator. The drugs will be filled in the syringes and the syringes handed over to on floor consultant anesthetist who are blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group BF (Experimental): hyperbaric Bupivacaine 10mg with fentanyl 10micrograms
  Interventions: Drug: Bupivacaine, fentanyl
- Group BD (Experimental): hyperbaric Bupivacaine 10 mg with dexmedetomidine5 micrograms
  Interventions: Drug: Bupivacaine, dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine, fentanyl — Group A: hyperbaric Bupivacaine 10mg with fentanyl 10micrograms,
  Arms: Group BF
Drug: Bupivacaine, dexmedetomidine — Group B: hyperbaric Bupivacaine 10 mg with dexmedetomidine5 micrograms
  Arms: Group BD

SUMMARY:
the primary objective of the study is to compare the onset and recovery times of sensory and motor blockade of the two study drugs intrathecally with low dose bupivacaine The secondary objectives of the study are to observe hemodynamics, side effects profile, and duration of postoperative analgesia

DETAILED DESCRIPTION:
The current study is undertaken to compare the effect of two drugs intrathecally.edexmedetomidine and fentanyl with a low dose of bupivacaine and assess the adequacy of the block, side effect profile and postoperative analgesia. The two drugs have been studied separately but the comparative data is scarcely available both at national and international level. A particular agent is a dexmedetomidine that has been introduced in the investiagator's setup for the first time so this research will be of great importance in adding its multiple uses other than being used as ICU and procedural sedation agent.

ELIGIBILITY:
Inclusion Criteria:

Term pregnancy Singleton ASA I and II, BMI <35, elective C/section

Exclusion Criteria:

patient refusal, contraindications to spinal anaesthesia. ASA III and IV, PIH Pre Eclampsia, allergic to Local Anesthetic, fetal anomalies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Time till T10 dermatome achieved (Sec) | Post operative initial hour
  Spinal block characteristics
Time of maximum bromage achieved (Sec) | Post operative initial hour
  Spinal block characteristics
Regression time to T10 dermatome (Min) | Post operative initial hour
  Spinal block characteristics
Time of complete motor recovery (Min) | Post operative initial hour
  Spinal block characteristics
Post-operative pain score | 1 hour
  VAS score indicate 0 no pain 10 severe pain. Pain score was noted down
Post-operative pain score | 2 hour
  VAS score indicate 0 no pain 10 severe pain. Pain score was noted down
Post-operative pain score | 3 hour
  VAS score indicate 0 no pain 10 severe pain. Pain score was noted down
Post-operative pain score | 4 hour
  VAS score indicate 0 no pain 10 severe pain. Pain score was noted down

SECONDARY OUTCOMES:
Nausea | 24 hours Post operative
  Sensation to throw out stomach contents
Vomiting | 24 hours Post operative
  Act of throwing out stomach contents through mouth
Pruritus | 24 hours Post operative
  Unpleasing sensation on the skin that provokes to scratch
Respiratory distress | 24 hours Post operative
  Difficulty in breathing
Shivering | 24 hours Post operative
  The act of shaking slightly and uncomfortably due to felling of cold temperature
Bradycardia | 24 hours Post operative
  Heat rate less than <60 bpm
Hypotension | 24 hours Post operative
  Decrease in BP greater than 20% of baseline

OTHER OUTCOMES:
Systolic Blood Pressure | Baseline
  Hemodynamics
Systolic Blood Pressure | Immediate after giving intrathecal injection and positoning
  Hemodynamics
Systolic Blood Pressure | at 5 minute
  Hemodynamics
SBP | at 10 minute
  Hemodynamics
Systolic Blood Pressure | at 15 minute
  Hemodynamics
Systolic Blood Pressure | at 20 minute
  Hemodynamics
Diastolic Blood Pressure | Baseline
  Hemodynamics
Diastolic Blood Pressure | Immediate after giving intrathecal injection and positoning
  Hemodynamics
Diastolic Blood Pressure | at 5 minute
  Hemodynamics
Diastolic Blood Pressure | at 10 minute
  Hemodynamics
Diastolic Blood Pressure | at 15 minute
  Hemodynamics
Diastolic Blood Pressure | at 20 minute
  Hemodynamics
Heart Rate | Baseline
  Hemodynamics
Heart Rate | Immediate after giving intrathecal injection and positoning
  Hemodynamics
Heart Rate | at 5 minute
  Hemodynamics
Heart Rate | at 10 minute
  Hemodynamics
Heart Rate | at 15 minute
  Hemodynamics
Heart Rate | at 20 minute
  Hemodynamics
oxygen saturation | Baseline
  Hemodynamics
oxygen saturation | Immediate after giving intrathecal injection and positoning
  Hemodynamics
oxygen saturation | at 5 minute
  Hemodynamics
oxygen saturation | at 10 minute
  Hemodynamics
oxygen saturation | at 15 minute
  Hemodynamics
oxygen saturation | at 20 minute
  Hemodynamics
respiratory rate | Baseline
  Hemodynamics
respiratory rate | Immediate after giving intrathecal injection and positoning
  Hemodynamics
respiratory rate | at 5 minute
  Hemodynamics
respiratory rate | at 10 minute
  Hemodynamics
respiratory rate | at 15 minute
  Hemodynamics
respiratory rate | at 20 minute
  Hemodynamics

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Civil Hospital Karachi, Karachi, Sindh
  - DUHS, Civil hospital Karachi (CHK), Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No